CLINICAL TRIAL: NCT07006779
Title: Effects of Music and Conversation on Pain and Anxiety Levels During Transrectal Ultrasound-Guided Prostate Biopsy: A Randomized-Controlled Prospective Study
Brief Title: Effects of Music and Conversation in Prostate Biopsy
Acronym: TRUS-BX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Volkan Selmi, Associate Professor, Bozok University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-KAEK-189_2021.05.05_08
Record Dates: First submitted 2025-05-15; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Prostate Neoplasms; Prostate Biopsy
Keywords: prostate biopsy; music; conversation; anxiety; pain
MeSH Terms: conditions — Prostatic Neoplasms; Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music intervention (Experimental): The patients who listened to music during procedure
  Interventions: Behavioral: Music intervention
- Conversation (Experimental): The patients who were involved into conversation during procedure
  Interventions: Behavioral: Conversation
- Control (No Intervention): The patients who were not involved into conversation or listened to music during procedure

INTERVENTIONS:
Behavioral: Music intervention — Engaging into conversation during procedure
  Other Names: Conversation
  Arms: Music intervention
Behavioral: Conversation — Engaging patients into conversation
  Arms: Conversation

SUMMARY:
The goal of this observational study is to learn about the effects of music and conversation on pain and anxiety levels during Transrectal Ultrasound-Guided Prostate Biopsy. The main question it aims to answer is:

Does music or conversation reduces the pain and anxiety levels of patients

DETAILED DESCRIPTION:
The patients who were scheduled to undergo TRUS-PBx were randomly assigned to one of three groups (n=30) via sealed envelope randomization method: the control group, the music group, and the conversation group.

Patients' sociodemographic data such as age, height, weight and body mass index were documented. The International Prostate Symptom Score (IPSS), PSA level and prostate volume of all patients was recorded before the procedure. Blood pressure and heart rate were checked before and after the procedure.

Patients completed the State-Trait Anxiety Inventory (STAI) test, which consists of 40 questions, with 20 questions each in the state and trait subscales, both before and after the procedure. Low scores indicated low anxiety levels, while high scores reflected higher anxiety levels. Also, anxiety and pain levels were assessed using a visual analog scale (VAS).

The procedure room was designed to minimize external disturbances (e.g., sound or noise). Prior to the biopsy, patients received detailed information according to their assigned group. In the music group, patient-selected music was played throughout the procedure. In the conversation group, discussions based on the patients' interests were initiated and continued during the procedure. In the control group, no additional interaction beyond the informational briefing was provided.

Post-procedure, patients were asked whether they would be willing to undergo the procedure again if necessary. Responses were categorized as "positive," "negative," or "abstained."

ELIGIBILITY:
Inclusion Criteria:

* pathological findings on Digital Rectal Examination
* PSA value greater than 2.5 ng/ml

Exclusion Criteria:

* psychiatric disorders,
* those who declined to participate,
* hearing or perceptual impairments,
* continuous analgesic use,
* history of prior prostate biopsy,
* prilocaine allergy were excluded.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male patients
Enrollment: 90 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale of Pain | Periprocedural
  pain levels were assessed using a visual analog scale (VAS), where a score of "0" indicated "no pain or anxiety," and a score of "10" represented "the most severe pain
Visual Analog Scale of Anxiety | Periprocedural
  Anxiety levels were assessed using a visual analog scale (VAS), where a score of "0" indicated "no pain or anxiety," and a score of "10" represented "the most severe anxiety
State-Trait Anxiety Inventory (STAI) test | Periprocedural
  State-Trait Anxiety Inventory (STAI) test, which consists of 40 questions, with 20 questions each in the state and trait subscales, both before and after the procedure. The test was scored using a 4-point Likert scale, with total scores ranging from 20 to 80. Low scores indicated low anxiety levels, while high scores reflected higher anxiety levels.

CONTACTS AND LOCATIONS:
Overall Officials: volkan selmi, Principal Investigator — Yozgat Bozok University
Locations (1):
- Yozgat Bozok University Research and Training Hospital, Yozgat, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chiu LP, Tung HH, Lin KC, Lai YW, Chiu YC, Chen SS, Chiu AW. Effectiveness of stress management in patients undergoing transrectal ultrasound-guided biopsy of the prostate. Patient Prefer Adherence. 2016 Feb 11;10:147-52. doi: 10.2147/PPA.S96991. eCollection 2016. PMID 26929606
- [Background] Cho SW, Choi HJ. Effect of Music on Reducing Anxiety for Patients Undergoing Transrectal Ultrasound-Guided Prostate Biopsies: Randomized Prospective Trial. Urol J. 2016 Apr 16;13(2):2612-4. PMID 27085561
- [Background] Chang YH, Oh TH, Lee JW, Park SC, Seo IY, Jeong HJ, Kwon WA. Listening to music during transrectal ultrasound-guided prostate biopsy decreases anxiety, pain and dissatisfaction in patients: a pilot randomized controlled trial. Urol Int. 2015;94(3):337-41. doi: 10.1159/000368420. Epub 2014 Dec 18. PMID 25531837
- [Derived] Selmi V, Taspinar MS, Caniklioglu M, Sari S, Akyuz M, Isikay L. Effects of music and conversation on pain and anxiety levels during transrectal ultrasound-guided prostate biopsy: a randomized-controlled prospective study. Sao Paulo Med J. 2025 Dec 15;144(1):e20253273. doi: 10.1590/1516-3180.2025.3273.28072025. eCollection 2025. PMID 41417393